CLINICAL TRIAL: NCT04855435
Title: A Phase I Multicentre, Open-label, Dose Escalation Study to Determine the Safety and Preliminary Efficacy of MBS8(1V270) Administered Intravenously to Cancer Patients With Advanced Solid Tumours
Brief Title: Safety and Preliminary Efficacy of MBS8(1V270) in Cancer Patients With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MonTa Biosciences ApS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBS8-101
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single arm, multinational, multicenter Phase I trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MBS8(1V270) (Experimental): Treatment arm (single arm study)
  Interventions: Drug: MBS8(1V270)

INTERVENTIONS:
Drug: MBS8(1V270) — The investigational medicinal product will be administered IV by infusion. Subjects will be treated in cycles.

SUMMARY:
The Phase I trial is planned to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of MBS8(1V270) in subjects with advanced solid tumours. The trial is designed to provide data for further clinical development of MBS8(1V270)

DETAILED DESCRIPTION:
This is a prospective, open-label, single arm, multinational, multicenter Phase I trial in subjects with advanced solid tumors.

The trial consists of two stages: Stage I is a dose escalation stage which will include up to eight cohorts with escalating doses of MBS8(1V270) to establish the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D). Stage II is an expansion phase in which safety and tolerability of MBS8(1V270) will be assessed at the recommended phase 2 dose established in Stage I of the trial.

The dose-escalation in stage 1 is based on the 1+2 design for the first cohort and on the 3+3 design for the following cohorts.

The investigational medicinal product is a TLR7 agonist and will be administered intravenously by infusion.

Subjects will be treated in cycles and the dose-limiting toxicity (DLT) observation period is 23 days.

Plasma cytokine levels will be assessed, and tumor biopsies will be taken and evaluated. Radiological tumor assessment by MRI or CT will be performed.

Safety will be evaluated by the incidence of adverse events (AEs), serious adverse events (SAEs), DLTs, and use of concomitant medications.

Anti-tumor activity of MBS8(1V270) will be evaluated via imaging using RECIST and iRECIST criteria, with iRECIST being the leading tumor evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years
2. Diagnosis of histologically- or cytologically-confirmed solid tumour that is advanced and with progression. No standard treatment exists, or the subject refuses standard treatment. Experimental immunotherapy appears as feasible exploratory treatment option as per investigator assessment.
3. Tumour lesion(s) accessible to serial biopsies.
4. Must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumour biopsies.
5. Measurable disease according to RECIST V1.1. Previously irradiated lesions are measurable if subsequent progression is documented.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. Life expectancy > 3 months as assessed by the investigator.
8. Adequate bone marrow, cardiopulmonary, renal and hepatic functions:

   * Haemoglobin ≥5.6 mmol/L (≥ 90 g/dL) (without transfusion or erythropoietin therapy within 4 weeks prior to therapy);
   * Neutrophils ≥1.5 x 109/L, without growth factor stimulation within 3 weeks prior to the blood test;
   * Platelet count ≥ 75 × 109/L;
   * Serum creatinine ≤ 1.25 times ULN or creatinine clearance ≥50 mL mL/min (by CKD-EPI formula);
   * Hepatic function: AST and ALT ≤ 2.5 x ULN; (5 × ULN in the case of liver metastases); bilirubin ≤ 1.5 × ULN except in case of Gilbert's disease and 2 × ULN in case of liver metastases.
9. All subjects of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must have a negative highly sensitive pregnancy test at screening (urine/serum) and agree to use highly effective method for contraception according to the European Union (EU) Clinical Trial Facilitation Group guidance from time of signing the informed consent form (ICF) until at least 120 days after the last administration of trial drug. The partners of subjects with childbearing potential must also apply contraceptive methods and are recommended not to donate sperm.
10. Ability to understand and sign the ICF.

Exclusion Criteria:

1. Has had biologic, hormonal, anti-neoplastic chemotherapy, or radiation therapy within 4 weeks prior to screening (6 weeks required for nitrosourea or mitomycin) except for medications with half-lives <5.5 days.
2. Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumour masses of large volume with close relation to the mayor airways where tumour necrosis may cause perforation or severe bleeding episodes. Primary or metastatic intestinal disease in situ where tumour necrosis may cause gastrointestinal perforation.
3. Use of investigational agent in the 4 weeks or 5 half-lives prior to first dose of MBS8(1V270), whichever is shortest.
4. Major surgical procedure within 14 days prior to the first trial drug dose.
5. Has a history of another primary malignancy, except for:

   * Malignancy treated with curative intent and with no known active disease within 2 years prior to first dose of MBS8(1V270).
   * Adequately treated non-invasive basal skin cancer or squamous cell skin carcinoma.
   * Adequately treated uterine cervical cancer stage 1B or less.
6. Treatment with systemic immunosuppressive medication (including but not limited to corticosteroids (>10 mg prednisone per day or equivalent, except topical or inhaled), cyclophosphamide, azathioprine, methotrexate, thalidomide, anti-IL-6 receptor agents and anti-TNFα agents) within 2 weeks prior to initiation of trial treatment, or anticipation of need for systemic immunosuppressive medication during trial treatment.
7. Treatment with androgen deprivation therapies such as luteinizing-hormone releasing hormone (LHRH) (gonadotropin-hormone releasing hormone [GnRH]) agonists within 2 weeks prior to initiation of trial treatment.
8. Ongoing immune-related adverse events (irAEs) and/or AEs ≥ Grade 2 not resolved from previous therapies except vitiligo, resolved atopy, limited psoriasis, stable neuropathy Grade 2, hair loss, and stable endocrinopathies with substitutive hormone therapy.
9. Has uncontrolled intercurrent or chronic illness, but not limited to, ongoing or active infection such as hepatitis B or C, human immunodeficiency virus (HIV), immune dysfunction such as autoimmune disease, psychiatric illness such as depression or suicidal tendency or social situations that would limit compliance with trial requirements.
10. Has active or history of immunologic-mediated disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome or Guillain-Barré syndrome.
11. Has clinically significant cardiac disease, including:

    * Known congestive heart failure Grade III or IV by the New York Heart Failure Association (see Appendix A);
    * Myocardial infarction within 6 months prior to signing the ICF;
    * Onset of unstable angina within 6 months prior to signing the ICF.
12. History of severe allergic episodes.
13. Known hypersensitivity to any component of MBS8(1V270).
14. Has a history of seizure disorders uncontrolled on medication.
15. Has a history of clinically significant coagulation or bleeding disorders or abnormalities.
16. Abnormal or clinically significant coagulation parameters at the discretion of the investigator, i.e.:

    * International Normalized Ratio (INR);
    * Activated Partial Thromboplastin Time (APTT). Subjects being treated with anticoagulants are excluded if the coagulation parameters are outside the therapeutic intervals as described in the Summary of Product Characteristics (SmPC) for the administered treatment.
17. Women of childbearing potential who deny remaining abstinent (refrain from heterosexual intercourse) or do not use a highly effective form of contraception that results in a failure rate of < 1% per year during the treatment period and up 120 days after the last trial drug administration.
18. Men of reproductive potential who deny to follow accepted contraception methods during treatment and up to 120 days after the last trial drug administration.
19. Pregnant or lactating women.
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, make administration of the trial drugs hazardous, or make it difficult to monitor adverse effects such that it is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has an autoimmune disorder requiring immune modulating treatment (>10 mg prednisone per day or equivalent, except topical or inhaled) during the last 2 years prior to first dose of MBS8(1V270).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 42 days
  Type and number of adverse events
Dose limiting toxicities | 23 days
  Dose limiting toxicities (DLTs) and the MTD for determination of RP2D of MBS8(1V270)
Safety related biomarkers | 23 days
  Plasma levels of safety related cytokines IL-6 and TNF-alpha wil be assessed

SECONDARY OUTCOMES:
Best overall response | 42 days
  Complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), unconfirmed (iUPD) and confirmed PD (iCPD), assessed according to Response Evaluation Criteria in Solid Tumours (RECIST) and immune RECIST (iRECIST
Progression free survival | 6 months
  The length of time a subject lives with the disease but without progression
Pharmacokinetic profile of drug substance | 22 days
  The plasma concentration time profile of MBS8(1V270) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer S Rohrberg, MD PhD, Principal Investigator — University Hospital of Denmark, Department of Oncology
Locations (5):
- Institut Jules Bordet, Anderlecht, Belgium
- Denmark (2):
  - University Hospital of Denmark, Department of Oncology, Copenhagen
  - Herlev and Gentofte Hospital, Center for Cancer Research, Herlev
- Spain (2):
  - Fundacion Instituto de Investigacion Sanitaria Fundacion Jimenez Diaz (FJD), Madrid
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid